CLINICAL TRIAL: NCT02855983
Title: Perforating Fat Injections for Plantar Fasciosis
Acronym: PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeffrey A. Gusenoff, MD, MD, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UPittsburgh_PRF
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Plantar Fascia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Fat grafting initially) (Experimental): A PATHWAY -
  Intervention: autologous fat grafting to the foot, occur first
  Fat graft study intervention procedure to occur first, next post-operative follow up visits (V1-V4). The Subject will after Month 6 (V4) crossover to Pathway B to complete Observation visits V1 (Month 2) and V2 (Month 6). After completion of V2 (Month 6), the subject will have completed study participation.
  Interventions: Procedure: Fat Grafting
- B (Standard of care initially) (Other): B PATHWAY -
  Intervention: standard of care (observation) for the first year, followed by autologous fat grafting to the foot
  Observation visit will occur first, next the subject will have two Observation visits V1 (Month 2) and V2 (Month 6). The subject will then crossover to Pathway A. The subject will be assessed by the PI his/her for continued study eligibility. Once the continued eligibility has been determined, the subject will have the interventional fat graft procedure and subsequent post-operative follow up visits (V1-V4). After completion of Post-op V4 (Month 6), the subject will have completed study participation.
  Interventions: Procedure: Fat Grafting

INTERVENTIONS:
Procedure: Fat Grafting — Grafting of autologous fat tissue is a minimally invasive surgical technique that starts with the harvest of fat tissue from the abdomen or thighs using liposuction through incisions less than 2mm in length. The lipoaspirate is then processed to concentrate the adipose fraction and reinjected into the graft site. This surgical procedure involves the immediate transplantation of a patient's own tissue in a single operative procedure.

SUMMARY:
The specific aim of this study is to determine whether perforating fat injections to the plantar fascia is a safe method to improve pain, quality of life, and reduce plantar fascia thickness for patients with chronic plantar fasciitis. We will also correlate the intrinsic fat properties of adipose stem cells (ie. growth factors) to the improvement in pain, quality of life, and plantar fascia thickness over time.

DETAILED DESCRIPTION:
Aim 1: Evaluate the safety of perforating fat injection into the plantar fascia in patients with chronic plantar fasciitis to improve pain, quality of life, and thickness of the fascia.

Rationale: Perforating fat injections have been shown to improve multiple scar and fibrotic conditions such as burn scar contracture, breast radiation injury, and Dupuytren's contracture of the hand. (5-7) It is thought that the perforations allow expansion of the tissues, and filling them with fat allows for a regenerative healing process, rather than an inflammatory scar healing process.

Hypothesis: Perforating fat injections into the chronically thickened plantar fascia is a safe method to improve pain, quality of life, and reduce tissue thickness.

Aim 2: Correlate intrinsic fat properties of lipoaspirate to improvement in function and plantar fascia thickness.

Rationale: Adipose tissue contains adipose derived stem cells. Various growth factors released from the stem cells may have a local effect on soft tissues (ie. VEGF). (8) These stem cells are thought to promote regenerative healing, rather than scar formation and may ultimately improve the thickness of the plantar fascia. (9-12) Hypothesis: Intrinsic fat properties of lipoaspirate (adipose stem cell characteristics) are closely correlated to the improvements in quality of life and thickness of the plantar fascia.

ELIGIBILITY:
Inclusion Criteria

Patients meeting the following criteria will be eligible to participate in the study:

1. Aged 18 years or older and able to provide informed consent
2. Subjects with a diagnosis of Plantar Fasciitis having heel pain that has not improved with splints, exercises or rountine standard of care treatment
3. Subjects must have a current relationship with their foot specialist managing the Plantar Fasciitis diagnosis.
4. Subjects must be 6 months post any surgical intervention to the affected foot
5. Subjects with a history of foot ulcer(s), the ulcer(s) must be healed with no recurrance for six months prior to consent to participate in this study.
6. Willing and able to comply with follow up examinations, including ultrasounds and radiographs
7. Subjects must be determined by the PI or a Co-Investigator to currently suffer from a diagnosis of chronic plantar fasciitis based on physician examination and foot evaluation.

Exclusion Criteria:

Patients with the following characteristics will be excluded from participating in the study:

1. Age less than 18 years
2. Inability to provide informed consent
3. Bilateral foot examination presents with open ulcerations, or diagnosis of osteomyelitis, non-healed fracture, neuropathy or tarsal tunnel syndrome.
4. Diabetics with a HgA1C >7
5. Current active and/or clinically significant infection identified anyway in the body, as demonstrated by physical assessment, laboratory findings, subject report and /or medical history.
6. Diagnosed with systemic or metastatic cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
7. Known coagulopathy
8. Systemic disease that would render the fat harvest and injection procedure, along with associated local anesthetic unsafe to the patient.
9. Any isssue that per the physician's determination would render the patient not appropriate to continue participation in the study (compliance, change in physical status, etc. )
10. Diagnosis of Pregnancy or the intent to of the participant to become pregnant during her participation in this study
11. Subjects with a diagnosis of Schizophrenia or Bipolar Disorder (Subjects who are found to be stable on medication and receive psychiatric clearance from a mental health professional could be eligible for study participation per the Physician's discretion).
12. Tobacco use: Last used anytime within 1 year, beginning and inclusive of date of study screening per subject report. Should the subject begin smoking during study participation, physician at time of notification in change in smoking status to determine subject's continued participation.
13. Morbid obesity: BMI>than or equal to 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Plantar fascia thickness | 6 months
  Assessed by ultrasound

SECONDARY OUTCOMES:
Local and systemic complications resulting from fat graft procedure | 6 months
  Including infection, fat necrosis, hematoma, seroma
Plantar foot pain | 6 months
  Assessed by validated foot pain questionnaries

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Gusenoff, MD, Principal Investigator — UPMC Department of Plastic Surgery
Locations (1):
- UPMC Plastic Surgery Aesthetic Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gusenoff BR, Minteer D, Gusenoff JA. Perforating Fat Injections for Chronic Plantar Fasciitis: A Randomized, Crossover Clinical Trial. Plast Reconstr Surg. 2022 Feb 1;149(2):297e-302e. doi: 10.1097/PRS.0000000000008765. PMID 35077429